CLINICAL TRIAL: NCT04656145
Title: The Efficacy of Chlorhexidine Gluconate Gel Dressing in Preventing Surgical Drain Site Infection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study team was not able to enroll eligible patients.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-01587
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Drain Site Complication
Keywords: Tegaderm

STUDY DESIGN:
Intervention Model Description: A paired study design will be used and subjects will serve as their own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Chlorhexidine Gluconate Gel Dressing (Experimental): All subjects are receiving two surgical drains during a single operative procedure. This arm will be randomized to receive the intervention.
  Interventions: Device: 3M™ Tegaderm™ CHG Chlorhexidine Gluconate I.V. Securement Dressing
- Standard of Care (No Intervention): All subjects are receiving two surgical drains during a single operative procedure. This arm will be randomized to received standard drain care - gauze (no intervention).

INTERVENTIONS:
Device: 3M™ Tegaderm™ CHG Chlorhexidine Gluconate I.V. Securement Dressing — On the day of the operation, after the procedure has concluded and the drains have been placed, the surgical drain site that has been randomized to be in the experimental group will receive the chlorhexidine gel dressing. The dressing will remain on the patient until the drain has been removed and the surgical site will be assessed for signs of infection.
  Arms: Chlorhexidine Gluconate Gel Dressing

SUMMARY:
This study aims to evaluate if the application of chlorhexidine gluconate dressing on surgical drain sites can decrease drain site infection vs the standard of care (dry, sterile gauze).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Receiving two surgical drains during one of the following types of operative procedures: breast reduction, breast augmentation, abdominoplasty, panniculectomy, brachioplasty, thigh lift, lower body lift, belt lipectomy, back latissimus dorsi reconstruction, bilateral breast reconstruction, or bilateral chest reconstruction. These drains may be in fairly close proximity to one another but they must emerge from different areas of the skin, that way they can be considered to be located in two different sites.

Exclusion Criteria:

1. Concurrent implantation of any foreign objects, such as a breast implant
2. Patients who receive postoperative antibiotics without a suspected or identified site of infection
3. Subjects allergic to or hypersensitive to chlorhexidine gluconate. Before enrolling in the study, patients will be asked about previous exposure to chlorhexidine products and about their allergies. Those with potential allergic or adverse reaction to chlorhexidine will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Erythema Measurement | Day 0, up to Month 6
  Drain site erythema will be measured with a ruler, in millimeters.
Number of participants in each category of skin induration (flat, soft, or firm) | up to Month 6
  2. Induration of skin will be measured by palpation of the skin around the drain by the clinician. This will be measured by assessing whether skin is flat, soft, or firm.
Change in distance between skin changes and normal looking skin | Day 0, up to Month 6
  Extent of skin changes is measured using a ruler, in millimeters, to calculate the distance between skin changes and normal looking skin.
Total amount of drainage from drain site | Up to Month 6
  Amount of drainage from drain site will be measured in cubic centimeters.
Number of participants who experience pain post-op | Up to Month 6
  5. Pain will be measured by asking patients if they experience pain (yes or no) when the clinician presses on the drain site.
Number of participants in each category of quality of drainage (serous, sanguineous, or purulent) | Day 0, up to Month 6
  Quality of drainage will be assessed by measuring thickness of drainage. Thickness of drainage will be measured as serous, sanguineous, or purulent.

SECONDARY OUTCOMES:
Number of participants displaying signs of wound infection | up to Month 6
  Measures of wound infection will be assessed by documenting any signs of cellulitis or abscess around the drain.
Number of participants displaying sterility of seroma | up to Month 6
  Sterility of seroma will be measured by assessing whether the serous collection of fluid has absence of infection.
Antibiotic prescription rate | up to Month 6
  This will be measured as the number of days that patients are prescribed antibiotics.
Number of participants displaying presence of hematoma | up to Month 6

CONTACTS AND LOCATIONS:
Overall Officials: David Chiu, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Thomas.Calahan@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.